CLINICAL TRIAL: NCT04782479
Title: The Effect of Practitioner's Hand Position on Tracheal Tube Movement While Removal of Stylet During Tracheal Intubation
Brief Title: Hand Position for Stylet Removal During Tracheal Intubation
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Associate professor, SMG-SNU Boramae Medical Center
Other Study IDs: 30-2018-18
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Manikin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- in the air: the position of the practitioner's hand holding the tube was placed in the air while the assistant pulling back the stylet.
  Interventions: Procedure: hand position
- on the cheek of a manikin: the position of the practitioner's hand holding the tube was placed on the cheek of a manikin while the assistant pulling back the stylet.
  Interventions: Procedure: hand position

INTERVENTIONS:
Procedure: hand position — For tracheal intubation with a stylet for a manikin, one time, the position of the hand holding the tube was placed in the air, and the other time, the position of the hand holding the tube was placed on the cheek of the patient, while the assistant pulling back the stylet.

SUMMARY:
Investigators compared the tube movement between two situations; the one was that the practitioner's hand holding the tracheal tube was placed in the air, and the other was that the hand was placed on the manikin's cheek, while two residents took the roles of the practitioner and the assistant in tracheal intubation with a stylet for a manikin.

DETAILED DESCRIPTION:
Residents who accepted spontaneous participation were randomly combined into teams of two each. For two residents in a team, each sequentially took on the role of a practitioner and once as an assistant for tracheal intubations by changing the position of the hand holding the tube; one time, the position of the hand holding the tube was placed in the air, and the other time, the position of the hand holding the tube was placed on the cheek of the manikin. For the assistant role, residents performed stylet removal with two hands. Investigators filmed a video of the tube movement while the assistant pulling up the stylet at 1/8x speed. While analyzing the captured videos, it was measured how much the tube held by the intubation practitioner went in front or how far back during the process of pulling the stylet.

ELIGIBILITY:
Inclusion Criteria:

* residents in the department of Anesthesia and Pain Medicine

Exclusion Criteria:

* refusal for participation

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Residents in the department of Anesthesia and Pain Medicine
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
tube movement distance | procedure (at the time when the assistant pulling back the stylet)
  tube movement distance in the process of pulling out the stylet by the assistant

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea